CLINICAL TRIAL: NCT03845634
Title: Validation of a Non-Motor Fluctuation Assessment Instrument (NoMoFA) for Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Assistive Technology Clinic, Canada (Other)
Collaborators: University of Cincinnati (Other); The Cleveland Clinic (Other); University Health Network, Toronto (Other); University of Michigan (Other); Rush University (Other); The Parkinson Study Group (Network)
Responsible Party: Sponsor
Other Study IDs: 10-27
Record Dates: First submitted 2019-02-07; First posted 2019-02-19 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Parkinson Disease
Keywords: Non-motor fluctuation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigators have developed a comprehensive questionnaire that assesses the presence of non-motor fluctuations (NMFs) in individuals with Parkinson's disease (PD). To date, 189 participants with PD have been assessed for preliminary data analysis prior to developing the penultimate version. At this time the objectives are to: (i) assess the scale's internal consistency and item-to-total correlations; (ii) assess test-retest reliability; (iii) use factor analysis and reliability measures to guide item reduction; (iv) assess construct validity; and (v) assess the scales ability to discriminate between static non-motor symptoms and non-motor symptoms which fluctuate (vi) estimate the relative distribution of cognitive, psychiatric, autonomic, sleep and sensory NMFs in PD patients with motor fluctuations and their impact on quality of life in Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Idiopathic Parkinson's Disease (according to the United Kingdom Parkinson's Disease Society Brain Bank clinical diagnostic criteria)
* Stage of symptoms is mild, moderate or severe as per the Hoehn & Yahr scale
* Have motor fluctuations
* Have non-motor fluctuations

Exclusion Criteria:

* Atypical Parkinsonism
* Lack of motor fluctuations
* Lack of English language proficiency in either subject or caregiver

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Individuals, both men and women, who have been diagnosed with idiopathic Parkinson's Disease and have motor and non-motor fluctuating symptoms are invited to participate in the study. To ensure a representative sample, subjects spanning the disease spectrum will be equally represented in terms of mild, moderate and advanced symptoms of PD.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2019-09-11 (Actual); Study Completion 2019-09-11 (Actual)

PRIMARY OUTCOMES:
Cronbach's Alpha | Baseline
  alpha 0 - 1.0
Item-to-total correlation | Baseline
  correlation -1.0 - 1.0
Inter-rater reliability | 1 week after Baseline
  kappa 0 - 1.0
Concurrent validity | Baseline
  correlation -1.0 - 1.0

CONTACTS AND LOCATIONS:
Overall Officials: Galit Kleiner, MD, Principal Investigator — Assistive Technology Clinic
Locations (1):
- Assistive Technology Clinic, Toronto, Ontario, Canada